CLINICAL TRIAL: NCT06870487
Title: An Open-Label Phase 1 Study to Evaluate PF-08046032 as Monotherapy and Part of Combination Therapy in Participants With Advanced Malignancies
Brief Title: A Study to Learn About the Study Medicine Called PF-08046032 in People With Advanced Cancers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C5911001; 2024-517756-35-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-02-24; First posted 2025-03-11 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Peripheral T Cell Lymphoma; Diffuse Large B-cell Lymphoma; Classical Hodgkin Lymphoma; Head and Neck Squamous Cell Carcinoma; Melanoma; Non-Small Cell Lung Cancer
Keywords: Solid tumors; Advanced Malignancies; Malignancies; Lung cancer; Skin cancer; Non-Hodgkin lymphoma; Hodgkin lymphoma; Advanced Cancers; Head and Neck Cancer; Metastatic Cancer; Blood Cancer
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, Large B-Cell, Diffuse; Squamous Cell Carcinoma of Head and Neck; Melanoma; Carcinoma, Non-Small-Cell Lung; Neoplasms; Lung Neoplasms; Skin Neoplasms; Lymphoma, Non-Hodgkin; Hodgkin Disease; Head and Neck Neoplasms; Neoplasm Metastasis; Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- PF-08046032 Monotherapy Dose Escalation (Experimental): PF-08046032 will be given as an intravenous (IV) infusion.
  Interventions: Drug: PF-08046032
- PF-08046032 + Sasanlimab Combination Safety Evaluation (Experimental): PF-08046032 will be given as an intravenous (IV) infusion and sasanlimab will be administered as a subcutaneous injection.
  Interventions: Drug: PF-08046032; Drug: Sasanlimab
- PF-08046032 + Sasanlimab Combination Expansion Cohort (Experimental): PF-08046032 will be given as an intravenous (IV) infusion and sasanlimab will be administered as a subcutaneous injection.
  Interventions: Drug: PF-08046032; Drug: Sasanlimab

INTERVENTIONS:
Drug: PF-08046032 — PF-08046032 will be administered intravenously (IV) infusion.
Drug: Sasanlimab — Sasanlimab will be administered as subcutaneous (SC) injection.
  Arms: PF-08046032 + Sasanlimab Combination Expansion Cohort; PF-08046032 + Sasanlimab Combination Safety Evaluation

SUMMARY:
The purpose of this study is to learn about the effects of a new study medicine called PF-08046032, when taken alone and when taken with another medicine called sasanlimab, for the treatment of advanced cancers. The effects are studied in adult participants with certain types of lymphomas or solid tumors that are advanced or metastatic (spread to other parts of the body).

The study has three parts:

* Part A will test PF-08046032 alone at increasing dose levels in participants with certain lymphomas (cancer that begins in cells of the immune system) and in participants with certain solid tumors whose disease has worsened on or after standard treatments.
* Part B will test PF-08046032 (at selected doses) and sasanlimab in participants with certain solid tumors, including those whose disease has worsened on or after standard treatments as well as participants before receiving standard treatments.
* Part C will further test the combination of PF-08046032 and sasanlimab in participants with specific types of solid tumors based on the results from Part A and Part B of the study.

All participants will receive the study drug PF-08046032. Only participants in Part B and Part C of the study will also receive sasanlimab. PF-08046032 will be given as an intravenous (IV) infusion, which means it will be injected directly into a vein. Sasanlimab will be given as a subcutaneous injection, which means it will be injected under the skin.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Histological or cytological diagnosis of metastatic or unresectable malignancy:

   * Part A1: Participants with lymphomas (cHL, PTCL, large B-cell lymphoma) who have progressed on/after standard therapies
   * Part A2: Participants with solid tumors (NSCLC, HNSCC, melanoma, or other limited tumor types) who have progressed on or following prior immune checkpoint inhibitor if indicated and available
   * Part B: Participants with solid tumors who have either progressed on/after prior immune checkpoint inhibitor, or who have not received prior immune checkpoint inhibitor therapy
   * Part C: Participants with selected tumor type who have not received systemic anticancer treatment for the tumor type (including prior immune checkpoint inhibitor
2. Measurable disease as defined by Lugano Classification for lymphomas or RECIST 1.1 for solid tumors
3. Able to provide tumor tissue(s) as defined by the protocol depending on the Part of the study at enrollment
4. ECOG Performance Status score 0 or 1

EXCLUSION CRITERIA:

1. Ongoing peripheral neuropathy
2. History of significant immune-mediated adverse event considered related to prior immune-modulatory therapy
3. Known or suspected active autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Part A and Part B: Number of participants with dose limiting toxicities (DLTs) in dose escalation | Day of first dose (Day 1) through the end of DLT Observation period (up to 28 days)
  DLT (any of the prespecified AEs that are attributable to study treatment(s), excluding toxicities clearly due to underlying disease or extraneous causes) rate estimated based on data from DLT-evaluable participants during the DLT evaluation period
All Parts: Number of participants with adverse events (AEs) | From first dose (Day 1) through up to 30 days after last dose of PF-08046032 or up to 90 days after last dose of sasanlimab
  AEs as characterized by type, frequency, severity (CTCAE v5), seriousness, and relationship to study drug(s)
All Parts: Frequency of dose modifications due to AEs | From first dose (Day 1) through up to 30 days after last dose of PF-08046032 or up to 90 days after last dose of sasanlimab
  Dose modifications such as dose delay, treatment interruptions, dose reducations, and treatment discontinuations due to AEs
All Parts: Number of participants with clinically significant lab abnormalities | From first dose (Day 1) through up to 30 days after last dose of PF-08046032 or up to 90 days after last dose of sasanlimab
  Lab abnormalities characterized by type, frequency, and severity (CTCAE v5)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) in Participants with Solid Tumors | Response assessments at baseline and every 8 to 12 weeks through time of disease progression, death, unacceptable toxicity, or through study completion (Approximately 3 Years)
  Based on investigator assessment, and defined as the proportion of participants who achieved best overall response of CR or PR according to RECIST 1.1
Duration of Response (DoR) in Participants with Solid Tumors | Time from first documented objective response to the date of first documented radiographic progression or death (Approximately 3 Years)
  Based on investigator assessment for participants with a confirmed objective response (CR or PR) only.
Progression-free survival (PFS) in Participants with Solid Tumors | Time from first dose (Day 1) to the date of first documented radiographic progression or death (Approximately 3 Years)
  Based on investigator assessment for tumor response/progression according to RECIST v1.1
Objective Response Rate (ORR) in participants with lymphomas based on Lugano Criteria | Response assessments at baseline and every 8 to 12 weeks through time of disease progression, death, unacceptable toxicity, or through study completion (Approximately 3 Years)
  Based on investigator assessment, and defined as the proportion of participants who achieved best overall response according to Lugano Criteria
Progression-free survival (PFS) in participants with lymphomas based on Lugano Criteria | Time from first dose (Day 1) to the date of first documented radiographic progression or death (Approximately 3 Years)
  Based on investigator assessment for tumor response/progression according to Lugano Response Classification Criteria
Duration of Response (DoR) in participants with lymphomas based on Lugano Criteria | Time from first documented objective response to the date of first documented radiographic progression or death (Approximately 3 Years)
  Based on investigator assessment for participants with a confirmed objective response only.
Complete Response Rate (CRR) in participants with lymphomas | Response assessments at baseline and every 8 to 12 weeks through time of disease progression, death, unacceptable toxicity, or through study completion (Approximately 3 Years)
  Based on investigator assessment, and defined as the proportion of participants who achieved best overall response of Complete Response (CR) according to Lugano Criteria
Duration of Complete Response (DCR) in participants with lymphomas | Time from first documented CR to the date of the first radiographic progression or death (Approximately 3 Years)
  Based on investigator assessment for participants with lymphoma with a confirmed objective response per Lugano Criteria only.
Part C only: Overall survival (OS) | Baseline through date of death or study completion, whichever occurs first (up to approximately 3 Years)
  OS is defined as time from first dose of study treatment to death due to any cause.
Part A2 only: Change from baseline of the number of CD25+ cells in tumor in response to PF-08046032 treatment | Baseline through about 7 weeks after first dose
  Change is evaluated from paired biopsies
Pharmacokinetics (PK): Serum Area Under the Curve (AUC) from Time Zero to Last Quantifiable Concentration (AUClast) | Cycle 1 and Cycle 2, and pre-and post-dosing on Day 1 of Cycle 3, 4, 6, 8, and every 4th cycle thereafter; and within approximately 30 days after last dose of study drug (each cycle is 28 days)
  AUClast of PF-08046032 as a monotherapy (Part A) and in combination with sasanlimab (Part B and Part C).
PK: Maximum Observed Serum Concentration (Cmax) | Cycle 1 and Cycle 2, and pre-and post-dosing on Day 1 of Cycle 3, 4, 6, 8, and every 4th cycle thereafter; and within approximately 30 days after last dose of study drug (each cycle is 28 days)
  Cmax of of PF-08046032 as a monotherapy (Part A) and in combination with sasanlimab (Part B and Part C).
PK: Half-life (t1/2) | Cycle 1 and Cycle 2, and pre-and post-dosing on Day 1 of Cycle 3, 4, 6, 8, and every 4th cycle thereafter; and within approximately 30 days after last dose of study drug (each cycle is 28 days)
  Half life of PF-08046032 as a monotherapy (Part A) and in combination with sasanlimab (Part B and Part C)
PK: Minimum observed serum concentration (Ctrough) | Cycle 1 and Cycle 2, and pre-and post-dosing on Day 1 of Cycle 3, 4, 6, 8, and every 4th cycle thereafter; and within approximately 30 days after last dose of study drug (each cycle is 28 days)
  Ctrough of PF-08046032 as a monotherapy (Part A) and in combination with sasanlimab (Part B and Part C)
PK: Time to Reach Maximum Observed Serum Concentration (Tmax) | Cycle 1 and Cycle 2, and pre-and post-dosing on Day 1 of Cycle 3, 4, 6, 8, and every 4th cycle thereafter; and within approximately 30 days after last dose of study drug (each cycle is 28 days)
  Tmax of PF-08046032 as a monotherapy (Part A) and in combination with sasanlimab (Part B and Part C)
Incidence of Anti-Drug Antibody (ADA): Immunogenicity of PF-08046032 as a single agent (Part A) and in combination with sasanlimab (Part B and Part C) | Pre-dose on Day 1 of Cycles 1-4, then cycle 6, 8, and every 4th cycle thereafter, and within approximately 30 days after last dose of study drug (each cycle is 28 days)
  Immunogenicity of PF-08046032 and in combination with sasanlimab

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (3):
  - NEXT Oncology, San Antonio, Texas
  - Fred Hutchinson Cancer Center., Seattle, Washington
  - University of Washington Medical Center- Montlake, Seattle, Washington
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona]
  - Hospital Universitario Fundación Jiménez Díaz, Madrid

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5911001